CLINICAL TRIAL: NCT04979611
Title: The Clinical Application of 68Ga-NOTA-exendin-4 PET/CT in Detecting Insulinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian11
Record Dates: First submitted 2021-07-27; First posted 2021-07-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Insulinoma
MeSH Terms: conditions — Insulinoma | interventions — 68Ga-NOTA-exendin-4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will undergo 68Ga-NOTA-exendin-4 PET/CT imaging (Other): A single dose of 37-111 Mega-Becquerel (MBq) 68Ga-NOTA-exendin-4 will be injected intravenously. PET/CT imaging will be performed at 30-60 min post-injection.Visual and semiquantitative method will be used to assess the PET/CT images.
  Interventions: Drug: 68Ga-NOTA-exendin-4

INTERVENTIONS:
Drug: 68Ga-NOTA-exendin-4 — A single dose of 37-111 Mega-Becquerel (MBq) 68Ga-NOTA-exendin-4 will be injected intravenously

SUMMARY:
The small insulinoma can not be detected by the CT or MRI. We use 68Ga-NOTA-exendin-4 positron emission tomography/computed tomography (PET/CT) to detect the insulinoma for the patient diagnosed with endogenous hyperinsulinemic hypoglycaemia. And the diagnostic value will be performed. A single dose of 37-111 Mega-Becquerel (MBq) 68Ga-NOTA-exendin-4 will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
The glucagon-like peptide-1 receptor (GLP-1R) is an emerging target due to its high expression in benign insulinomas. 68Ga-NOTA-exendin-4 is an optimal probe targeting GLP-1R. The clinical use of 68Ga-NOTA-exendin-4 PET/CT in detecting insulinomas will be evaluated. And the comparation between PET diagnostic value and CT / MRI will be done.

ELIGIBILITY:
Inclusion Criteria:

* 1.age ≥6 years old 2.Patients with hypoglycaemia 3.Endogenous hyperinsulinemic hypoglycaemia 4.Enhanced CT or MRI within 1 month 5.Signed written consent

Exclusion Criteria:

* 1. Breast feeding 2.Pregnancy or the wish to become pregnant within 6 months 3.Renal function: serum creatinine during 41-73umol/L 4.Any medical condition may significantly interfere with study compliance; 5.Known allergy

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV) | From right after tracer injection to 1-hours post-injection
  Determination of SUV for detected lesions and discernible organs of 68Ga-NODAGA-JR11 and 68Ga-DOTATATE Standard uptake value (SUV) of the lesion will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China